CLINICAL TRIAL: NCT05874934
Title: Endoscopic Drainage of Presumed Resectable Perihilar Cholangiocarcinoma Using an Intrahepatic Plastic Stent With Retrieval String; a Pilot Study (CHORDA-II-pilot)
Brief Title: Endoscopic Drainage of Presumed Resectable pCCA Using an Intrahepatic Plastic Stent With Retrieval String
Acronym: CHORDA-II-p
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Rogier P. Voermans, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.0249; NL83570.018.22 (Other: CCMO)
Record Dates: First submitted 2023-02-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: Biliary drainage; Intrahepatic plastic stent with retrieval string; Presumed resectable perihilar cholangiocarcinoma
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intrahepatic plastic biliary stent with retrieval string
  Interventions: Device: Intrahepatic biliary stent with retrieval string

INTERVENTIONS:
Device: Intrahepatic biliary stent with retrieval string — Plastic biliary stent with 3-0 nylon (ethilon) thread tied to the distal end of the stent through the existing sidehole.

SUMMARY:
Prospective pilot study to assess the feasibility and efficacy of intrahepatic plastic biliary stents with a retrieval string in patients with presumed resectable perihilar cholangiocarcinoma requiring biliary drainage of the future liver remnant.

DETAILED DESCRIPTION:
Background: Pre-operative biliary drainage is advised to treat obstructive jaundice and optimize the clinical condition of patients with presumed resectable perihilar cholangiocarcinoma who are expected to be eligible for major liver resection. However, stent related complications such as cholangitis (37%) and stent dysfunction (19%) occur frequently. Creating the need for numerous re-interventions, re-admissions, delay of diagnostic work-up and potential surgery. Biliary drainage could be optimized by the use of a navel design short fully covered self-expanding metal stent (FCSEMS) which is currently examined in the CHORDA-pilot study. However, FCSEMS placement is not feasible in an considerable number of cases, in these patients the use of a plastic stent with a retrieval string could be beneficial over standard plastic stent placement, which makes removal possible although the stent does not reach into the duodenum.

Objective: To explore feasibility and efficacy of endoscopic drainage of patients with presumed perihilar cholangiocarcinoma eligible for major liver resection using a plastic stent with a retrieval string.

Study population: Patients with presumed perihilar cholangiocarcinoma that are judged eligible for major liver resection and require endoscopic biliary drainage of the future liver remnant.

lntervention: Endoscopic drainage of the future liver remnant using a plastic biliary stent with retrieval string (diameter 7 or 1 0Fr).

Primary outcome: Number of severe drainage related complications between inclusion and exploratory laparotomy. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever comes first.

Secondary study parameters/outcome of the study (if applicable):

Secondary outcomes: technical and therapeutic success of biliary drainage, individual components of primary endpoints and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Capable of providing written and oral informed consent.
* Presumed perihilar cholangiocarcinoma.
* Biliary obstruction in the future liver remnant.
* Drainage naïve patients: total bilirubin >50 umol/L
* Patients with previous endobiliary drainage procedures: persistently rising total bilirubin >50 umol/L (i.e. no stent placed or insufficient draining stent) or persistent biliary dilatation in the future liver remnant on imaging (i.e. previous stent placed in contralateral side of the liver).

Exclusion Criteria:

* Incompletely recovered from any side effects of previous biliary drainage procedures. Patients are required to be off antibiotic treatment for at least 5 days.
* Any contra-indication for major liver surgery (e.g. ECOG/WHO score ≥3).
* Technical contra-indications for endobiliary drainage (e.g. previous gastrojejunostomy).
* Distance between stricture and sphincter less than 2 cm.
* Refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Severe adverse events between inclusion and exploratory laparotomy | Between inclusion and surgery. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever
  Number of severe drainage related complications between inclusion and exploratory laparotomy. Severe complications are defined as any complication leading to additional invasive interventions, (extended) hospitalization, or death.

SECONDARY OUTCOMES:
The separate incidence of preoperative cholangitis between inclusion and exploratory laparotomy | Between inclusion and surgery. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever
  Number of patients who experience preoperative cholangitis.
Technical success of intervention | Between inclusion and surgery. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever
  The number of drainage procedures required to achieve technical success.
Therapeutic success of intervention within 14 days | 14 days
  The number of patients who with therapeutic success, defined as normal caliber bile ducts in the future liver remnant on ultrasound examination and a decrease in total bilirubin concentration of at least 20% at day 7 relative to the concentration at baseline.
Number of drainage procedures between inclusion and exploratory laparotomy | Between inclusion and surgery. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever
  The total number of drainage procedures that involved (attempted) stent (re-)placement.
Bilirubin levels after 7 and 14 days | 14 days
  Interval bilirubin decrease at 7 days and 14 days after biliary drainage relative to the bilirubin level at inclusion.
Cancellation of surgery | Between inclusion and surgery. In patients who will not undergo exploratory laparotomy, the number of drainage-related complications will be measured until 7 days after the decision to cancel exploratory laparotomy or 90 days after inclusion, whichever
  The number of patients with rescheduled or cancelled laparotomy due to severe drainage-related complications.
Quality of life after 7 days. | 7 days
  EORTC Quality of Life Questionnaire 30 (EORTC QLQ-30), the EORTC QLQ module for CCA and gallbladder cancer (EORTC QLQ-BIL21), and the EuroQol 5D (EQ-5D-5L). Scoring according to module, higher score means better outcome.
Quality of life after 28 days. | 28 days
  EORTC Quality of Life Questionnaire (EORTC QLQ-30 incl BIL-21 module and EQ-5D-5L). Scoring according to module, higher score means better outcome.
Quality of life after 90 days. | 90 days
  EORTC Quality of Life Questionnaire (EORTC QLQ-30 incl BIL-21 module and EQ-5D-5L). Scoring according to module, higher score means better outcome.
Postoperative morbidity | 30 days after surgery
  EORTC Quality of Life Questionnaire (EORTC QLQ-30 incl BIL-21 module and EQ-5D-5L). Scoring according to module, higher score means better outcome.
Postoperative mortality | 30 days after surgery
  Number of patients experiencing postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Rogier P. Voermans, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Pending